CLINICAL TRIAL: NCT04627441
Title: A Pilot Study of the Characterization of Transcutaneous and Epidural Spinal Stimulation for Enabling Motor Function in Humans With Motor Complete Paraplegia
Brief Title: Transcutaneous and Epidural Stimulation in SCI
Acronym: Service-Line
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-related delays and insufficient funding.
Sponsor: Kristin Zhao, PhD (Other)
Responsible Party: Sponsor-Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-006477
Record Dates: First submitted 2020-10-15; First posted 2020-11-13 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Paraplegia, Spinal; Paraplegia, Complete; Paraplegia; Traumatic
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TESS-EES (Experimental): Transcutaneous Electrical Spinal Stimulation (TESS), used during the first month of training sessions, followed by Epidural Electrical Stimulation (EES) during the final 6-month training period.
  Interventions: Device: Transcutaneous spinal cord stimulator; Device: Epidural spinal cord stimulator system

INTERVENTIONS:
Device: Transcutaneous spinal cord stimulator — DS8R Electrical Stimulator For Human Research
Device: Epidural spinal cord stimulator system — Spectra WaveWriter Epidural Spinal Cord Stimulator System with CoverEdge 32 Electrode Surgical Lead

SUMMARY:
The study seeks to improve the scientific understanding of how two electrical stimulation techniques, one which delivers electricity to the skin surface over the spine (transcutaneous electrical spinal stimulation [TESS]) and another which is implanted onto the dura mater of the spinal cord (epidural electrical stimulation [EES]), facilitate spinal circuitry to enable function after SCI.

DETAILED DESCRIPTION:
The study will compare motor activity and clinical outcomes over the course of TESS and EES in combination with physical rehabilitation.

The primary outcome data collected will be used to characterize and compare spinal sensorimotor activity in muscles below the level of injury during TESS and EES-enabled motor tasks in persons with chronic motor complete paralysis of the lower extremities due to traumatic SCI. Furthermore, data collected will be used as a proof of concept that TESS can be used to determine recovery of function during EES-enabled motor tasks. Following exposure to each stimulation intervention, data collection will include changes to spasticity, body composition, metabolic variables, and spinal imaging to assess the effect of either TESS or EES stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury due to trauma located between the seventh cervical (C7) and tenth thoracic vertebrae (T10)
* American Spinal Injury Association grading scale of A or B (4 each of A and B) below the level of SCI
* Intact spinal reflexes below the level of SCI
* At least 1-year post-SCI
* At least 22 years of age
* Willing to use medically acceptable methods of contraception, if female and of child-bearing potential

Exclusion Criteria:

* Currently a prison inmate, or awaiting trial, related to criminal activity
* Pregnancy at the time of enrollment
* Dual energy x-ray absorptiometry (DEXA) t-score <-3.5 at spine and femur head
* History of chronic and/or treatment resistant urinary tract infection
* Unhealed decubitus ulcer
* Unhealed skeletal fracture
* Untreated clinical diagnosis of depression
* Presence of joint contractures or an Ashworth spasticity score of 4
* Active anti-spasticity medication regimen within 3 months prior to study enrollment
* Presence of transcranial magnetic stimulation-evoked potentials in leg muscles
* Undergoing, or planning to undergo, diathermy treatment
* Active participation in another interventional clinical trial
* Presence of conditions or disorders which require MRI monitoring
* A history of coagulopathy or other significant cardiac or medical risk factors for surgery
* Current use of a ventilator
* Clinically diagnosed cardiopulmonary complications such as chronic obstructive pulmonary disease, cardiac failure, or heart arrhythmia that contraindicate changes in body position such as supine-to-sit-to-stand activities, prolonged standing, or stepping
* Mass > 113 kg (250 pounds)
* History of frequent hypotension characterized by light headedness, or loss of consciousness
* History of frequent hypertension characterized by headache, or bradycardia
* History of frequent, severe, autonomic dysreflexia
* Any illness or condition which, based on the research team's assessment, will compromise with the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during this study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-16 (Estimated); Primary Completion 2025-12-16 (Estimated); Study Completion 2025-12-16 (Estimated)

PRIMARY OUTCOMES:
Kinematics | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of joint angles, measured in degrees.
Electromyography | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of electrical activity at major muscle groups below the level of injury.
Foot pressure | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of foot pressure through shoe-insole pressure sensors.
Overground ambulation [as appropriate to the subject] (1) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in overground mobility as measured by the Modified 6 Minute Walk Test. Trainers will assess the distance in meters which the subject can cover in 6 minutes, with a greater distance characterizing better overground mobility.
Overground ambulation [as appropriate to the subject] (2) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in walking impairment as measured by the Walking Index for Spinal Cord Injury. Trainers will assess overall level of impairment, ranging from most severe impairment (0) to least severe impairment (20), based on the use of devices, braces, and physical assistance of one or more persons.
Somatosensory evoked potentials | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of change in conduction in the peripheral nerves, cervical and lumbosacral spinal cord, deep brain structures, and sensory cortex, through surface electrodes.
Transcranial magnetic stimulation motor evoked potentials | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of stimulus intensity required to elicit muscle responses in muscle groups known to elicit optimal motor evoked potential responses, both above and below the level of injury.
Monosynaptic spinal reflex testing | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of stimulation intensity H and F wave thresholds and maximal responses through surface electrodes.
Trunk stability | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of trunk stability using the modified functional reach test (mFRT).
Injury severity: American Spinal Injury Association (ASIA) Impairment Scale | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of impairment of sensory and motor functions using the American Spinal Injury Association Impairment Scale. Individuals are classified from A" (complete spinal cord injury) to "E" (normal function). 28 dermatomes and 10 key muscles are assessed bilaterally. Results are summed to produce overall sensory and motor scores and are used in combination with evaluation of anal sensory and motor function as a basis for the determination of ASIA classification. Sensory scores are rated 0 (sensation absent) to 2 (normal), bilaterally for each of 28 dermatomes. Muscle function is rated 0 (total paralysis) to 5 (active movement, full range of motion against significant resistance) for each myotome. Upper Extremity Motor Subscores and Lower Extremity Motor Subscores are each scored from 0 to 50; the ASIA Motor Score is scored from 0 to 100. The presence of anal sensation and voluntary anal contraction are assessed as a yes/no.

SECONDARY OUTCOMES:
Spasticity | Baseline, End of TESS, Start of EES, End month 6 EES
  Change in measurements of spasticity using the Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET). Answers to qualitative questions are rated from -3 to +3, with a higher positive number indicating more helpful symptoms, and a lower negative number indicating more problematic symptoms. Scores are totaled for a score which categorizes the overall positive or negative impact of a subject's spasticity symptoms.
Bone mineral density | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement by dual-energy x-ray absorptiometry (DEXA) of change in bone mineral content and bone density.
Body composition - body fat mass | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement by dual-energy x-ray absorptiometry (DEXA) of change in regional and total body fat mass.
Body composition - lean mass | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement by dual-energy x-ray absorptiometry (DEXA) of change in regional and total lean mass.
Body composition - android and gynoid fat percentage | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement by dual-energy x-ray absorptiometry (DEXA) of change in regional and total android and gynoid fat percentage.
Body composition - bone mass | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement by dual-energy x-ray absorptiometry (DEXA) of change in regional and total bone mass.
Metabolics - CBC | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in complete blood count with differential.
Metabolics - glucose | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in fasting glucose value.
Metabolics - total cholesterol | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in total cholesterol value.
Metabolics - HDL cholesterol | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in HDL cholesterol value.
Metabolics - calculated LDL cholesterol | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in calculated LDL cholesterol value.
Metabolics - triglycerides | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in triglycerides value.
Metabolics - non-HDL cholesterol | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in non-HDL cholesterol value.
Neurostimulator array location and migration | Start of EES, End month 6 EES
  Evaluation of current array location via CT.
Patient-reported bowel function (1) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in bowel function using the Neurogenic Bowel Dysfunction Score. Answers to qualitative questions are rated from 0 to 5, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes severity of neurogenic bowel symptoms.
Patient-reported bowel function (2) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in bowel function using the International Spinal Cord Injury Bowel Function Basic Data Set (v2.0). Answers to qualitative questions are rated from 0 to 13, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes neurogenic bowel dysfunction.
Patient-reported bladder function (1) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in bladder function using the Neurogenic Bladder Symptom Score. Answers to qualitative questions are rated from 0 to 5, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes severity of neurogenic bladder symptoms.
Patient-reported bladder function (2) | Baseline, End of TESS, Start of EES, End month 6 EES
  Assessment of change in bowel function using the International Spinal Cord Injury Urodynamic Basic Data Set. Data from various urodynamic variables are aggregated into a single-page format for an abstract overview of bladder dysfunction.
Male patient-reported sexual function (1) | Baseline, End of TESS, Start of EES, End month 6 EES
  Assessment of change in sexual function using the International Spinal Cord Injury Male Sexual Function Basic Data Set (v2.0). Data from various male sexual function variables are aggregated into a single-page format for an abstract overview of male sexual dysfunction.
Male patient-reported sexual function (2) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in erectile dysfunction using the Sexual Health Inventory for Men (SHIM). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better erectile function, and totaled for a score which categorizes severity of erectile dysfunction.
Male patient-reported sexual function (3) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in erectile dysfunction using the International Index for Erectile Function (IIEF). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better erectile function, and totaled for a score which categorizes severity of erectile dysfunction.
Female patient-reported sexual function (1) | Baseline, End of TESS, Start of EES, End month 6 EES
  Assessment of change in sexual function using the International Spinal Cord Injury Female Sexual and Reproductive Function Basic Data Set (v2.0). Data from various female sexual and reproductive function variables are aggregated into a single-page format for an abstract overview of female sexual and reproductive dysfunction.
Female patient-reported sexual function (2) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in sexual function using the Female Sexual Function Index (FSFI). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better sexual function, and totaled for a score which categorizes severity of sexual dysfunction.

OTHER OUTCOMES:
Volitional movement (1) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in volitional movement through recordings of training time in minutes.
Volitional movement (2) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in volitional movement through recordings body weight support measured as a percentage of total body weight supported.
Volitional movement (3) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of change in volitional movement through recordings of speed in miles per hour.
Volitional movement (4) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in volitional movement through recordings of assistive devices used.
Volitional movement (5) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in volitional movement through recordings of stimulator electrode location.
Volitional movement (6) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in volitional movement through recordings of stimulator intensity, measured in milliamps per volt.
Volitional movement (7) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurements of changes in volitional movement through recordings of stimulator frequency measured in Hertz.
Volitional movement (8) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in volitional movement through recordings of pulse width, measured in microseconds.
Overground ambulation [as appropriate to the subject] (1) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in severity of walking impairment as measured by the Walking Index for Spinal Cord Injury (WISCI II). Trainers combine the type of assistive device(s) used, use or no use of orthotic braces, number of persons assisting ambulation, and distance subject is able to walk (up to 10 meters), into a single score ranging from 0 to 20, with a lower number indicating more severe impairment.
Overground ambulation [as appropriate to the subject] (2) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in overground mobility as measured by the Modified 6 Minute Walk Test. Trainers will assess the distance in meters which the subject can cover in 6 minutes, with a greater distance characterizing better overground mobility.
Overground ambulation [as appropriate to the subject] (3) | Baseline, End of TESS, Start of EES, End month 6 EES
  Measurement of changes in overground mobility as measured by the Modified Timed Up and Go test. Trainers will assess the time it takes, in minutes and seconds, for the subject to stand from a chair, move out to a 3 meter distance, return to the chair and sit down. Less time will characterize better overground mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D. Zhao, Ph.D., Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials